CLINICAL TRIAL: NCT04589052
Title: Identification of Anxiety and Depression in Adolescents/Young Adults (AYA) With Cancer
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Julie Germann, Associate Professor of Psychiatry, University of Texas Southwestern Medical Center
Other Study IDs: STU-2019-1203
Record Dates: First submitted 2020-04-21; First posted 2020-10-19 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Cancer; Depression, Anxiety
MeSH Terms: conditions — Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, multisite (but all within the UTSW IRB), observational study assessing the relationship of hope to anxiety and depression, QoL, and social support over time in the first year after cancer diagnosis or relapse in AYA (ages 15-29 years of age).

DETAILED DESCRIPTION:
The principal investigators' ongoing work suggests hope is a target for intervention to improve quality of life (QoL) and reduce anxiety and depression (A/D) among adolescents/young adults (AYA). No study to the investigators' knowledge has evaluated the promising impact of hope interventions in AYA cancer patients. To address this gap, the investigators will expand the investigators' prior research on hope, A/D, and QoL to AYA receiving care across three diverse healthcare systems.

Patients will be approached for participation within 3 months of their initial/relapse cancer diagnosis. Eligible patients (and the parent/caregiver for minor patients) will be approached in a private area of the clinic or hospital room to explain the research aims and informed consent process. After obtaining informed consent/assent (from parents if patients are under 18, from AYA if patient is 18 or older), participants (patients) will utilize an iPad to complete measures via Redcap.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults (15-17, 18-29 years of age, respectively) with a new or relapse diagnosis of a malignancy
* Patients will include those being followed (treatment or observational) for any malignant disorder at Children's Medical Center, UT Southwestern Medical Center, or Parkland Health and Hospital Systems
* Patients whose native language is Spanish or English are eligible to participate
* Patients may have any life expectancy
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients with clinically apparent cognitive disabilities which would preclude understanding and completion of measures.
* Patients with significant medical issues such as delirium which preclude their ability to consent and complete initial measures

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents and young adults newly diagnosed as having a malignancy
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of a multi-site, multiple time-point psychosocial study for AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  * Hypothesis a: Greater than 50% of eligible patients will enroll and complete at least two time points in the study.
  * Hypothesis b: Enrollment and study completion rates will differ by site, with the site with the most psychosocial risk (low socioeconomic status as measured by insurance type (private, public, uninsured)) having the lowest enrollment and study completion rates.
  * Hypothesis c: Enrollment and study completion rates will differ by treatment type. Those receiving treatment that has the most frequent clinic/hospital visits (as measured by chemotherapy versus radiation only/surgery only) will have the highest completion rates.

SECONDARY OUTCOMES:
Correlation between hope and quality of life (QoL) in AYA cancer patients | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: Hope (as measured by Snyder's (1991) Hope Scale, higher scores indicate higher hope) will be positively correlated to QoL (Pediatric Quality of Life Inventory 3.0 - Cancer Module, PedsQL, Varni, 2002; higher scores indicate better quality of life)
Correlation between hope and social support (SS) in AYA cancer patients | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: Hope (as measured by Snyder's (1991) Hope Scale, higher scores indicate higher hope) will be positively correlated to SS (Multidimensional Perceived Social Support Scale (MPSSS; Zimet, Dahlem, Zimet, Farley, 1988); higher scores indicate higher social support)
Correlation between hope and anxiety and depression (A/D) in AYA cancer patients | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: Hope (as measured by Snyder's (1991) Hope Scale, higher scores indicate higher hope) will be inversely correlated to A/D (The Four-Item Patient Health Questionnaire for Anxiety and Depression (PHQ-4; Kroenke, Spitzer, Williams, & Löwe, B. (2009); higher scores indicate greater symptoms of anxiety/depression).
Determine the impact of medical factors (treatment) on hope in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: Medical severity (type of treatment (chemotherapy, surgery, radiation) will be inversely related to hope (The Hope Scale (Snyder et al., 1991); higher scores indicate greater hope)
Determine the impact of medical factors (treatment) on QoL in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: Medical severity (type of treatment (chemotherapy, surgery, radiation) will be inversely related to QoL (Pediatric Quality of Life Inventory 3.0 - Cancer Module (Varni, Burwinkle, Katz, Meeske, & Dickinson, 2002); higher scores indicate greater quality of life)
Determine the impact of medical factors (treatment) on AD in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: Medical severity (type of treatment (chemotherapy, surgery, radiation) will be positively related to A/D (The Four-Item Patient Health Questionnaire for Anxiety and Depression (PHQ-4; Kroenke, Spitzer, Williams, & Löwe, B. (2009); higher scores indicate greater symptoms of anxiety/depression)
Determine the impact of medical factors (treatment) on SS in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: Medical severity (type of treatment (chemotherapy, surgery, radiation) will be inversely related to SS (Multidimensional Perceived Social Support Scale (MPSSS; Zimet, Dahlem, Zimet, Farley, 1988); higher scores indicate greater social support).
Determine the impact of socieconomic status on hope in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: SES as indicated by insurance status will be inversely related to hope (The Hope Scale (Snyder et al., 1991); higher scores indicate greater hope)
Determine the impact of socieconomic status on QOL in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: SES as indicated by insurance status will be inversely related to QoL (Pediatric Quality of Life Inventory 3.0 - Cancer Module (Varni, Burwinkle, Katz, Meeske, & Dickinson, 2002); higher scores indicate greater quality of life)
Determine the impact of socieconomic status on AD in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: SES as indicated by insurance status will be positively related to A/D (The Four-Item Patient Health Questionnaire for Anxiety and Depression (PHQ-4; Kroenke, Spitzer, Williams, & Löwe, B. (2009); higher scores indicate greater symptoms of anxiety/depression)
Determine the impact of socieconomic status on SS in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: SES as indicated by insurance status will be inversely related to SS (Multidimensional Perceived Social Support Scale (MPSSS; Zimet, Dahlem, Zimet, Farley, 1988); higher scores indicate greater social support).
Determine the impact sex on hope in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: sex will be inversely related to hope (The Hope Scale (Snyder et al., 1991); higher scores indicate greater hope)
Determine the impact sex on QoL in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: sex will be inversely related to QoL (Pediatric Quality of Life Inventory 3.0 - Cancer Module (Varni, Burwinkle, Katz, Meeske, & Dickinson, 2002); higher scores indicate greater quality of life)
Determine the impact sex on AD in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: sex will be positively related to A/D (The Four-Item Patient Health Questionnaire for Anxiety and Depression (PHQ-4; Kroenke, Spitzer, Williams, & Löwe, B. (2009); higher scores indicate greater symptoms of anxiety/depression)
Determine the impact sex on SS in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: sex will be inversely related to SS (Multidimensional Perceived Social Support Scale (MPSSS; Zimet, Dahlem, Zimet, Farley, 1988); higher scores indicate greater social support).
Determine the impact of age on hope in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: age will be inversely related to hope (The Hope Scale (Snyder et al., 1991); higher scores indicate greater hope)
Determine the impact of age on QoL in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: age will be inversely related to QoL (Pediatric Quality of Life Inventory 3.0 - Cancer Module (Varni, Burwinkle, Katz, Meeske, & Dickinson, 2002); higher scores indicate greater quality of life)
Determine the impact of age on AD in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: age will be positively related to A/D (The Four-Item Patient Health Questionnaire for Anxiety and Depression (PHQ-4; Kroenke, Spitzer, Williams, & Löwe, B. (2009); higher scores indicate greater symptoms of anxiety/depression)
Determine the impact of age on SS in AYA with cancer | up to 12 months (+/- one 4 weeks) following enrollment
  - Hypothesis a: age will be inversely related to SS (Multidimensional Perceived Social Support Scale (MPSSS; Zimet, Dahlem, Zimet, Farley, 1988); higher scores indicate greater social support).

CONTACTS AND LOCATIONS:
Overall Officials: Julie Germann, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center / Children's Medical Center, Dallas, Texas, United States